CLINICAL TRIAL: NCT01909492
Title: Measurement of Relaxin in the Serum and Cerebrospinal Fluid of Subjects With and Without the Relapsing Form of Multiple Sclerosis
Brief Title: Measurement of Relaxin Peptide in Multiple Sclerosis (MS)
Status: Completed | Type: Observational
Sponsor: Providence Health & Services (Other)
Collaborators: Microstein, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 13-089B
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Results first posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; MS; Relaxin
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Blood Specimen Collection; Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patients will provide blood and cerebrospinal fluid for use in this research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Group 1 will consist of 10 subjects with suspected MS, who have had a clinical attack within the last 12 weeks, have at least one gadolinium-enhancing lesion on brain or spinal cord MRI taken within the prior 4 weeks, and for which they have not received any immunomodulating or immunosuppressant medication. Patients will have a blood draw to provide serum and a CSF will be obtained through a lumbar puncture.
  Interventions: Procedure: Blood Draw; Procedure: Lumbar Puncture
- Group 2: Group 2 will consist of 10 subjects with clinically stable definite MS, with no evidence of clinical relapse for at least the past 12 weeks, and have no gadolinium enhancing lesions on MRI in the prior 4 weeks. These subjects will fulfill the Revised (2010) McDonald's Criteria for the Diagnosis of MS. Patients will have a blood draw to provide serum and a CSF will be obtained through a lumbar puncture.
  Interventions: Procedure: Blood Draw; Procedure: Lumbar Puncture
- Group 3: Group 3 will consist of 10 subjects without evidence of inflammatory systemic or inflammatory central nervous system disease, who require CSF removal for some other cause, such treatment of benign intracranial hypertension or as part of the procedure for insertion of an intrathecal medication delivery system. Patients will have a blood draw to provide serum and a CSF will be obtained through a lumbar puncture.
  Interventions: Procedure: Blood Draw; Procedure: Lumbar Puncture

INTERVENTIONS:
Procedure: Blood Draw — Patients will provide a serum sample for research.
Procedure: Lumbar Puncture — Patients will have a lumbar puncture to obtain CSF.
  Other Names: Spinal tap; LP

SUMMARY:
This study will evaluate relaxin (RLX) levels in patients with multiple sclerosis.

DETAILED DESCRIPTION:
The goal of this study is to obtain baseline information on serum and cerebrospinal fluid (CSF) relaxin levels in patients with MS, as well as to further study RXFP-1 receptor binding affinity for RLX in patients with active and clinically stable MS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with suspected MS, who have had a clinical attack within the last 12 weeks, have at least one gadolinium-enhancing lesion on brain or spinal cord MRI taken within the prior 4 weeks, and for which they have not received any immunomodulating or immunosuppressant medication.
* Subjects with clinically stable definite MS, with no evidence of clinical relapse for at least the past 12 weeks, and have no gadolinium enhancing lesions on MRI in the prior 4 weeks. These subjects will fulfill the Revised (2010) McDonald's Criteria for the Diagnosis of MS.
* Subjects without evidence of inflammatory systemic or inflammatory central nervous system disease, who require CSF removal for some other cause, such treatment of benign intracranial hypertension or as part of the procedure for insertion of an intrathecal medication delivery system.

Exclusion Criteria:

- Pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with suspected MS undergoing a lumbar puncture for diagnosis, patients with stable MS willing to participate in the study, and patients without MS having a lumbar puncture as part of their non-MS disease management will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-09-20 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Cohan, MD, PhD, Principal Investigator — Providence Brain & Spine Institute, Providence Health & Services
Locations (1):
- Providence MS Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 8 | 10 | 9 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Relaxin (RLX) Levels
Description: There is no information available on what serum and CSF levels of RLX are observed in patients with active versus stable relapsing MS, how these values compare to that found in human volunteers without MS or other inflammatory diseases, and whether RLX functions normally in subjects with active or stable MS. RLX2 concentrations were expressed as picomoles per milliliter (pmol/mL) of serum or CSF.
Time Frame: During diagnostic LP
Measure: Number; unit: pmol/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 10 | 10 | 10
pmol/mL
  RLX2 concentration level solely in serum | NA — Serum and CSF samples obtained from all of the volunteers, with or without a diagnosis of MS, failed to reveal RLX2 measurable above or equal to the LLD for the employed assay. | NA — Serum and CSF samples obtained from all of the volunteers, with or without a diagnosis of MS, failed to reveal RLX2 measurable above or equal to the LLD for the employed assay. | NA — Serum and CSF samples obtained from all of the volunteers, with or without a diagnosis of MS, failed to reveal RLX2 measurable above or equal to the LLD for the employed assay.
  RLX2 concentration level solely in the CSF | NA — Serum and CSF samples obtained from all of the volunteers, with or without a diagnosis of MS, failed to reveal RLX2 measurable above or equal to the LLD for the employed assay. | NA — Serum and CSF samples obtained from all of the volunteers, with or without a diagnosis of MS, failed to reveal RLX2 measurable above or equal to the LLD for the employed assay. | NA — Serum and CSF samples obtained from all of the volunteers, with or without a diagnosis of MS, failed to reveal RLX2 measurable above or equal to the LLD for the employed assay.

ADVERSE EVENTS:
Time Frame: Approximately 24 hours after the LP procedure research staff will contact the patient by phone to discuss any symptoms or serious adverse events
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 9/10 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=10) | Group 2 (N=10) | Group 3 (N=10)
Generalized soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache/Headaches (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Low back tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache secondary to lumbar puncture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Anxiety secondary to lumbar puncture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Soreness at LP procedure site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Headache post procedure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
mild upper respiratory congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache post LP (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain secondary to lumbar puncture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Headache (localized to back of head) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lightheaded (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Weakness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Minor back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Shortcomings of this study that may have confounded the data or its interpretation include the small sample sizes, no diagnostic group exceeding 10 volunteers, sample acquisition and handling and/or damage in shipment to Quanterix laboratories.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT01909492/Prot_SAP_000.pdf